CLINICAL TRIAL: NCT06049758
Title: D2 Versus D3 Dissection in Laparoscopic Right Hemicolectomy In Right Cancer Colon Patients: A Randomized Controlled Trial
Brief Title: D2 Versus D3 Dissection in Laparoscopic Right Hemicolectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Principal Investigator, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlexUni_D2D3
Record Dates: First submitted 2023-06-12; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Blood Loss; Intensive Care; Anastomotic Leakage; Lymph Node Disease; Survival; Blood Transfusion
MeSH Terms: conditions — Hemorrhage; Anastomotic Leak | interventions — Methods; Enoxaparin; Levofloxacin; Congresses as Topic

STUDY DESIGN:
Intervention Model Description: randomized controlled trial, single-blind, with randomized block randomization
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic hemicolectomy with Complete Mesocolic Excision (Active Comparator): Patients will have laparoscopic hemicolectomy with Complete Mesocolic Excision, D3 lymph node dissection.
  Interventions: Procedure: LAPAROSCOPIC RIGHT HEMICOLECTOMY procedure (intervention); Drug: Enoxaparin 40 Mg/0.4 mL Injectable Solution; Drug: Levofloxacin 500mg
- Conventional laparoscopic right hemicolectomy (Active Comparator): Patients will have conventional laparoscopic right hemicolectomy with D2 lymph node dissection.
  Interventions: Drug: Enoxaparin 40 Mg/0.4 mL Injectable Solution; Drug: Levofloxacin 500mg; Procedure: LAPAROSCOPIC RIGHT HEMICOLECTOMY procedure (Conventional)

INTERVENTIONS:
Procedure: LAPAROSCOPIC RIGHT HEMICOLECTOMY procedure (intervention) — Patients with right-side colon cancer (caecum, ascending, or hepatic flexure); were diagnosed by CT entero-colonography, colonoscopy, and biopsy who undergo laparoscopic right hemicolectomy
  Arms: Laparoscopic hemicolectomy with Complete Mesocolic Excision
Drug: Enoxaparin 40 Mg/0.4 mL Injectable Solution — Enoxaparin sodium 40 mg subcutaneous injection will be administered 12 hours before the operation
Drug: Levofloxacin 500mg — Levofloxacin 500 mg intravenous injection will be administered 1 hour before the operation.
Procedure: LAPAROSCOPIC RIGHT HEMICOLECTOMY procedure (Conventional) — Patients with right-side colon cancer (caecum, ascending, or hepatic flexure); were diagnosed by CT entero-colonography, colonoscopy, and biopsy who undergo laparoscopic right hemicolectomy
  Arms: Conventional laparoscopic right hemicolectomy

SUMMARY:
Evaluating the differences between D2 and D3 lymphadenectomy in laparoscopic right hemicolectomy in patients with right cancer colon post-operative outcome, intra-operative blood transfusion, post-operative ICU admission, anastomotic leakage, lymph node harvesting in the final specimen, and six months follow up and overall survival time after 5-years

DETAILED DESCRIPTION:
Surgical Technique and Preparation Enoxaparin sodium 40 mg subcutaneous injection will be administered 12 hours before the operation, and Levofloxacin 500 mg intravenous injection will be administered 1 hour before the operation.

Procedures will be performed under general anesthesia.

Group A:

Location of trocars and surgeons:

The patient will be placed in the Trendelenburg position and tilt to the left, with the surgeon standing between the patient's legs, the camera operator standing on the patient's left side, the assistant standing on the right of the camera operator, and the scrub nurse standing on the patient's right side.

1. A 30º-angled scope placed through port from an incision 5 cm below the umbilicus and two cm to the left to get an adequate view.
2. A 10-mm trocar will be introduced 10 cm below the umbilicus for the surgeon's right hand
3. 5-mm McBurney's point port will be placed for the left-hand instrument.
4. An additional two 5-mm trocars will be placed at the opposite McBurney's point and the left subcostal position for the assistant to retract and display the colon and mesocolon.

Surgical approach group A Tumor presence is confirmed by visual and tactile examination after thorough abdominal exploration.

First, the omentum will be turned up to the upper quadrant and the small intestine will be moved to the left, and the ileocecal junction and the root of the mesentery will be exposed.

Then, the appendix or caecum will be grasped and retracted in a lateral, anterior, and cranial direction by the assistant's left hand; the last ileal loop will be grasped and elevated by the assistant's right hand with an atraumatic bowel grasping forceps. Therefore, the mesentery root will be put under tension by this suspension.

Retrocolic dissection by cutting the peritoneum along the line between the right mesocolon and retroperitoneum) along the caudal aspect of the root and 1 cm above the right iliac vessels, as the entry for separation of the fusion fascial space between the visceral and parietal peritoneum (toldt fascia).

The right Toldt's fascia will be dissected and expanded medial to the periphery of the superior mesenteric vein (SMV), cranial to the pancreas head, and lateral to the ascending colon.

The posterior paries of ileocolic vessels (ICVs), right colic vessels (RCVs), and Henle's of gastro-colic trunk will be exposed.

Second, the mesocolon between the ICV and SMV will be dissected safely, and the ICV, RCV, and right gastroepiploic vessels as well as the right branch of the middle colic vessel will be divided and ligated easily because of the separated retroperitoneal space.

The lymph nodes along the SMV and SMA will be dissected using a caudal-to-cranial approach.

The greater omentum will be dissected for full mobilization of the mesocolon containing 10 cm of normal colon distal to the lesion followed by complete mobilization of the lateral attachments of the ascending colon.

Using laparoscopic stapler division of the transverse colon 10 cm distal to the tumor and last 20 cm of the ileum.

Anastomosis:

A functional side-to-side ileocolic intracorporeal anastomosis between the ileum and the transverse colon will be performed by liner stapler then closing enterostomy using 3/0 vicryl.

Extraction:

of the specimen through a midline or pfannenstiel incision; the incision length will be about 5-6 cm. A drain will be placed in the pelvis.

Group B:

Location of trocars and surgeons:

The patient will be placed in the Trendelenburg position and tilt to the left; the main surgeon and camera operator will stand to the left of the patient and the second assistant will be between the legs of the patient.

1. A 30º-angled scope placed through port from an incision through the umbilicus.
2. A 10-mm trocar will be introduced at left lumbar region for right working hand.
3. A 5-mm trocar will be introduced at left iliac region for left working hand.
4. A 10-mm trocar will be introduced at suprapubic for the assistant.
5. A 5-mm trocar will be introduced at right sub costal for the assistant. Surgical approach group B First, the pedicle of ileocolic vessels will be identified and the mesocolon will be dissected between the pedicle and the periphery of the Superior mesenteric vein（SMV）to expose the second portion of the duodenum.

The ileocolic vessels will then cut at their roots. The ascending mesocolon will be separated from the retroperitoneal tissues, duodenum, and pancreatic head up to the hepatocolic ligament cranially.

The important detail in this procedure is the wide separation between the pancreatic head and the transverse mesocolon. Using laparoscopic stapler division of the transverse colon 10 cm distal to the tumor and the last 20 cm of the ileum.

Anastomosis:

A liner stapler will perform a functional side-to-side ileocolic intracorporeal anastomosis between the ileum and the transverse colon, then closing enterostomy using 3/0 vicryl.

Extraction:

The specimen will go through a midline or Pfannenstiel incision; the length of the incision will be about 5-6 cm. A drain will be placed in the pelvis. This approach is the medial-to-lateral (MtL) approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with right-side colon cancer (caecum, ascending, or hepatic flexure)
* Diagnosed by CT entero-colonography
* Diagnosed by colonoscopy
* Diagnosed by biopsy.

Exclusion Criteria:

* Emergency surgery (obstruction, perforation with generalized peritonitis),
* Metastatic tumor diagnosed
* ASA score of IV or higher
* Need for more than one surgical procedure
* Conversion to open surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2026-01-02 (Estimated); Study Completion 2030-01-02 (Estimated)

PRIMARY OUTCOMES:
Number of blood units needed | during the intervention/procedure/surgery
  Guided by hemoglobine levels during surgery
Number of post-operative ICU admission | immediately after the intervention/procedure/surgery
  Incidence of ICU admission after surgery
Number of anastomotic leakage | Within 30 days post-operative
  incidence of anastomotic leakage
Number of lymph node harvesting in the final specimen | 6 months post-operative
  incidence of lymph node
Number of postoperative outcomes | 6 months post-operative
  the medical condition from the patient

SECONDARY OUTCOMES:
Overall survival time after 5-years | 5 years post-operative
  Survival analysis

CONTACTS AND LOCATIONS:
Overall Officials: Medhat Mohamed Anwar Hamed, Prof, Principal Investigator — Alexandria University
Locations (1):
- The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The analysis will be performed on a blinded dataset after completing the medical/scientific review. All protocol violations will be identified and resolved, and the dataset will be declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com), handled according to Good Clinical Practice guidelines, Data Protection Directive certificate, and complied with Title 21 CFR Part 11. Furthermore, the data centers where all the research data will be stored are certified according to ISO27001, ISO9001, and Dutch NEN7510.
  Can be asked by the contact person
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: whole study period
Access Criteria: ask contact person

REFERENCES:
- [Background] Colon Cancer Laparoscopic or Open Resection Study Group; Buunen M, Veldkamp R, Hop WC, Kuhry E, Jeekel J, Haglind E, Pahlman L, Cuesta MA, Msika S, Morino M, Lacy A, Bonjer HJ. Survival after laparoscopic surgery versus open surgery for colon cancer: long-term outcome of a randomised clinical trial. Lancet Oncol. 2009 Jan;10(1):44-52. doi: 10.1016/S1470-2045(08)70310-3. Epub 2008 Dec 13. PMID 19071061
- [Background] Pigazzi A, Hellan M, Ewing DR, Paz BI, Ballantyne GH. Laparoscopic medial-to-lateral colon dissection: how and why. J Gastrointest Surg. 2007 Jun;11(6):778-82. doi: 10.1007/s11605-007-0120-4. PMID 17562120
- [Background] Adamina M, Manwaring ML, Park KJ, Delaney CP. Laparoscopic complete mesocolic excision for right colon cancer. Surg Endosc. 2012 Oct;26(10):2976-80. doi: 10.1007/s00464-012-2294-4. Epub 2012 May 2. PMID 22549374
- [Background] Benz S, Tam Y, Tannapfel A, Stricker I. The uncinate process first approach: a novel technique for laparoscopic right hemicolectomy with complete mesocolic excision. Surg Endosc. 2016 May;30(5):1930-7. doi: 10.1007/s00464-015-4417-1. Epub 2015 Jul 21. PMID 26194254
- [Background] Watanabe T, Itabashi M, Shimada Y, Tanaka S, Ito Y, Ajioka Y, Hamaguchi T, Hyodo I, Igarashi M, Ishida H, Ishiguro M, Kanemitsu Y, Kokudo N, Muro K, Ochiai A, Oguchi M, Ohkura Y, Saito Y, Sakai Y, Ueno H, Yoshino T, Fujimori T, Koinuma N, Morita T, Nishimura G, Sakata Y, Takahashi K, Takiuchi H, Tsuruta O, Yamaguchi T, Yoshida M, Yamaguchi N, Kotake K, Sugihara K; Japanese Society for Cancer of the Colon and Rectum. Japanese Society for Cancer of the Colon and Rectum (JSCCR) guidelines 2010 for the treatment of colorectal cancer. Int J Clin Oncol. 2012 Feb;17(1):1-29. doi: 10.1007/s10147-011-0315-2. Epub 2011 Oct 15. PMID 22002491
- [Background] Kobayashi H, West NP, Takahashi K, Perrakis A, Weber K, Hohenberger W, Quirke P, Sugihara K. Quality of surgery for stage III colon cancer: comparison between England, Germany, and Japan. Ann Surg Oncol. 2014 Jun;21 Suppl 3:S398-404. doi: 10.1245/s10434-014-3578-9. Epub 2014 Feb 25. PMID 24566862
- [Background] Willaert W, Mareel M, Van De Putte D, Van Nieuwenhove Y, Pattyn P, Ceelen W. Lymphatic spread, nodal count and the extent of lymphadenectomy in cancer of the colon. Cancer Treat Rev. 2014 Apr;40(3):405-13. doi: 10.1016/j.ctrv.2013.09.013. Epub 2013 Sep 25. PMID 24126120
- [Background] Lee SD, Lim SB. D3 lymphadenectomy using a medial to lateral approach for curable right-sided colon cancer. Int J Colorectal Dis. 2009 Mar;24(3):295-300. doi: 10.1007/s00384-008-0597-7. Epub 2008 Oct 21. PMID 18941759
- [Background] Storli KE, Sondenaa K, Furnes B, Nesvik I, Gudlaugsson E, Bukholm I, Eide GE. Short term results of complete (D3) vs. standard (D2) mesenteric excision in colon cancer shows improved outcome of complete mesenteric excision in patients with TNM stages I-II. Tech Coloproctol. 2014 Jun;18(6):557-64. doi: 10.1007/s10151-013-1100-1. Epub 2013 Dec 20. PMID 24357446
- [Background] Bertelsen CA, Kirkegaard-Klitbo A, Nielsen M, Leotta SM, Daisuke F, Gogenur I. Pattern of Colon Cancer Lymph Node Metastases in Patients Undergoing Central Mesocolic Lymph Node Excision: A Systematic Review. Dis Colon Rectum. 2016 Dec;59(12):1209-1221. doi: 10.1097/DCR.0000000000000658. PMID 27824707
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245